CLINICAL TRIAL: NCT01309347
Title: Evaluation of the Development of an Advanced, Conformable Prosthetic Socket, Study I
Status: Completed | Type: Observational
Sponsor: Infoscitex Corporation (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kristen Leroy, Group Leader, Biomedical Devices, Infoscitex Corporation
Other Study IDs: IST-1288 Study I; W81XWH-07-C-0094 (Other Grant/Funding Number: US Army / TATRC)
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Evaluation of a New Prosthetic Socket Liner Material.
Keywords: prosthetic socket, residual limb volume fluctuation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is obtain prosthetist's feedback on the novel conformable socket material developed by Infoscitex, and determine if it is a viable alternative to current prosthetic socket liners. During this task, the research team will travel to the prosthetists locations to have them evaluate the socket system by examining the material and providing their professional opinions and feedback with regard to comfort and fit for the amputee, its ease of use, and breathability.

DETAILED DESCRIPTION:
Modern prosthetics have improved significantly with regards to control and functionality, but the fit of the residual limb within a prosthetic socket is a primary concern for many amputees. A poor fit can lead to skin irritation, tissue breakdown, and pain. The volume of the residual limb of an amputee changes throughout the course of a day and throughout the year. Volume fluctuation within the socket can lead to issues for the amputee, including decreased comfort, increased shear forces, increased pressure on bony prominences, as well as a poor gait pattern. An uncomfortable or non-performing socket/residual limb interface decreases user compliance with the prosthetic and therefore decreases the activity level of amputees who want to remain active in their civilian and military lives.

The investigators are developing a multilayered socket that takes advantage of a novel braided material for strength and passive conformability with thin layers dedicated to wearer comfort. This new socket provides ultimate fit for improvement in the performance of the prosthesis. The socket adapts itself to the changing physical shape of the residual limb as the prosthesis is worn. The adaptation is a natural result of the material properties, so is done passively and in real time. The materials are lightweight, breathable, and ultrasound transparent, allowing the prosthetic to function in a variety of environments.

This study will be undertaken to have six prosthetists evaluate the material, where they will be asked to complete a questionnaire and give their opinions regarding the material. This will inform design changes for the material.

ELIGIBILITY:
Inclusion Criteria:

* prosthetists who are active professionals and have clients (or have had clients in the past 6 months)

Exclusion Criteria:

* prosthetists who are not American Board for Certification of Orthotics and Prosthetics certified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study will be conducted at one prosthetic fabrication facility.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen LeRoy, Principal Investigator — Infoscitex Corporation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States